CLINICAL TRIAL: NCT06330207
Title: An Emergency Department (ED) Provider Centered Intervention for Non-Traumatic Dental Condition Management (NTDC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202301471; K99DE031723 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-03-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-04

CONDITIONS: Emergency Department Visit; Odontalgia
Keywords: non-traumatic dental conditions; emergency department; opioid; antibiotic
MeSH Terms: conditions — Toothache; Emergencies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): ED providers who will test the clinical decision support tool when prescribing for patients with non traumatic dental conditions
  Interventions: Behavioral: Clinical decision support tool

INTERVENTIONS:
Behavioral: Clinical decision support tool — The intervention involves two strategies. The first strategy is education where at baseline participants will complete the one-hour online Smiles for Life oral health educational module on acute dental problems, which includes NTDC management. This module can be completed in multiple sessions. Providers will be asked to share the certificate of completion that is provided to them via the website by passing a post knowledge test. The second strategy is CDST. Providers who completed NTDC module certificate will pilot test the CDST which is an algorithm that walks the ED provider thru patient's signs and symptoms and identifies guideline-recommended treatments available in the ED.

SUMMARY:
The overall objective of this proposal is to understand the barriers and facilitators to non-traumatic dental condition (NTDC) management in the emergency department (ED) through quantitative and qualitative methods. The first aim will determine the national variation in NTDC prescribing in the ED and subsequent ED/urgent care revisits and hospitalizations within 30-days of an index ED visit. Using national electronic health records and integrated claims datasets and a random effects model, we will identify factors associated with prescribing for NTDC and variation at the patient, provider, hospital and state levels. The second aim identifies ED providers' perceived barriers and facilitators to the management of NTDC in the ED. Using individual in depth interviews, ED providers (physicians, advanced practice providers) will identify the facilitators and barriers to management and prescribing for NTDC in the ED.

ELIGIBILITY:
Inclusion Criteria:

* ED providers (physicians, nurse practitioners, physician assistants)
* Working full-time in the ED

Exclusion Criteria:

* Part-time ED providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability and feasibility | at baseline, and up to 6 months
  Using qualitative methods, we will evaluate acceptability using the Theoretical Framework for Acceptability (TFA). Participants will complete a structured interview about acceptability at baseline and after 6 months of use, which should be sufficient time for providers to treat 5-10 patients for whom the tool is applicable. We pre-specify the criteria to define feasibility using criteria adapted from the NIH. Monthly during the trial, providers will answer feasibility surveys, using a web-based tool (i.e, RedCap) distributed via email. We will follow up with non-responders via text message, phone, or in-person. Providers will be offered a $5 gift card per survey as an incentive. To fully assess the impact of our intervention, we pre-specified a high retention rate as key to inform feasibility and effectiveness of future large-scale trials. We will consider successful implementation if >50% of providers intend to continue using the NTDC CDST postpilot.

SECONDARY OUTCOMES:
Prescribing behavior | at baseline, and up to 6 months
  For each participant, we will collect baseline antibiotic and opioid prescribing rates (per ED visit) for NTDC 6 months prior to the intervention from the EHR using the UPMC data analytics tool. All ED prescriptions in our system are created electronically, allowing precise capture of actual provider behavior. We will compare opioid and antibiotic prescribing for NTDC by providers before and after the intervention. To control for secular changes in prescribing, we will compare prescribing by participants during the same 6 months to prescribing by UPMC peers who did not receive the intervention.

OTHER OUTCOMES:
Pilot trial outcomes | up to 6 months post intervention
  We will develop good clinical practices to enhance the rigor and reproducibility of the research. This includes development of documentation, informed consent procedures, data collection tools, regulatory reporting, and monitoring procedures. In this pilot, we will evaluate possible outcome measures to quantify changes in ED provider NTDC management behavior. Qualitative and quantitative data generated will inform any necessary refinements to the intervention. This will provide a platform for larger evaluation to assess the effectiveness of our intervention for improving NTDC management in the ED.